CLINICAL TRIAL: NCT01042301
Title: Profiling of Original Cellular and Humoral Biomarkers of Type 1 Diabetes
Acronym: Lymphoscreen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BRD07/5-A
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Cordocentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Long-term type 1 diabetic patients (Experimental): Long-term type 1 diabetic patients
  Interventions: Other: Blood samplings
- control patients (Active Comparator): control patients
  Interventions: Other: Blood samplings
- diabetic and transplanted patients (Experimental): diabetic and transplanted patients
  Interventions: Other: Blood samplings
- subjects with high risk for diabetes (Experimental): subjects with high risk for diabetes
  Interventions: Other: Blood samplings
- patients with recent type 1 diabetes (Experimental): patients with recent type 1 diabetes
  Interventions: Other: Blood samplings
- patients with Latent Autoimmune Diabetes (Experimental): patients with Latent Autoimmune Diabetes
  Interventions: Other: Blood samplings

INTERVENTIONS:
Other: Blood samplings

SUMMARY:
The "Lymphoscreen" study aims to characterize precisely (phenotypes/cytokines/functions) CD8+ T cell responses in type 1 Diabetes to identify biomarkers of the disease. Such markers are needed for refine type 1 Diabetes diagnosis/prognostic, and to design new therapeutic approaches targeting autoreactive CD8+ T cells. An original approach using DNA immunization of humanized mice allowed us to identify relevant CD8 epitopes derived from GAD65 and IA-2 beta cell autoantigens. The aims are: (i) identifying exhaustively epitopes recognized by autoreactive CD8+ T lymphocytes in type 1 Diabetes and following islet or pancreas graft in humans; (ii) identifying pathogenic CD8+ T cell patterns or profiles related to type 1 Diabetes pathogenesis and evolution; (iii) correlating CD8+ autoreactive T cell responses and autoantibody responses to new cellular (such as CD4+ T cells or peripheral cell miRNA) or humoral markers of the disease (such as serum miRNA).

ELIGIBILITY:
Inclusion criteria:

* at least, 50 patients with "recent" type 1 diabetes,
* 30 patients with long-term type 1 diabetes,
* 10 patients with Latent Autoimmune Diabetes,
* 10 subjects with a risk for diabetes,
* 20 type 1 diabetic patients with pancreatic graft or Langerhans islet graft.
* 50 healthy subjects paired to HLA class I and to the age

Those subjects have to respect the following criteria :

* Age from 7 to 70 -Caucasian
* Affiliated to a national insurance scheme
* Written informed consent obtained For children, written informed consent is required from the two parents.

Non-inclusion criteria :

* Age strictly inferior to 7 or strictly superior to 70 years old
* Pregnancy
* Secondary diabetes
* No written informed consent

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Identification and characterization of new CD8+ T lymphocytes related to type 1 diabetes and its evolution (2009-2012) | 3 years

SECONDARY OUTCOMES:
Identification and characterization of new profiles of humoral and cellular markers (including T cell reactivity and miRNA) related to type 1 diabetes (2010-2014). | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Chaillous, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France